CLINICAL TRIAL: NCT01180829
Title: Pilot Study of Text Message Brief Interventions for Problem Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Health Canada (Other Government)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 088/2010
Record Dates: First submitted 2010-08-09; First posted 2010-08-12 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control condition (No Intervention): No interventions text messages sent
- Personalized feedback text messages (Experimental): A series of 12 text messages, each of which contains one personalized feedback item about the person's drinking
  Interventions: Behavioral: Personalized feedback text messages
- Consciousness raising text message (Experimental): A series of 12 text messages, each of which contains text designed to get the person to think about his or her drinking
  Interventions: Behavioral: Consciousness raising text messages

INTERVENTIONS:
Behavioral: Personalized feedback text messages — A series of 12 text messages, each of which contains one personalized feedback item about the person's drinking.
  Arms: Personalized feedback text messages
Behavioral: Consciousness raising text messages — A series of 12 text messages, each of which consists of an item designed to get the person to think about his or her drinking
  Arms: Consciousness raising text message

SUMMARY:
This study will provide a pilot test of two different text message interventions for problem drinkers. Participants will be recruited using a general population telephone survey. Participants in a control group (who will not receive text messages) will be compared to participants who receive one of two different types of text message packages (12 text messages sent once per week in each) - a series of personalized feedback text messages or a series of consciousness raising test messages (i.e., messages that keep the thought of cutting down on their drinking in the participants' mind). Participants in the three different conditions will be followed-up in three months time to assess changes in drinking. It is predicted that participants who receive either of the text message packages will report reduced drinking as compared to those participants in the control condition who do not receive any text messages.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Ontario
* 19 years of age or over
* Have consumed alcohol in the one month prior to the telephone survey.
* A score of 8 or over on the Alcohol Use Disorders Identification Test (AUDIT)
* Are willing to participate in follow-up at three months

Exclusion Criteria:

•None

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of drinks in a typical week | Three months

SECONDARY OUTCOMES:
Frequency of consumption | Three months
usual number of drinks per occasion | Three months
Frequency of consuming 5 or more drinks on one occasion | three months
highest number of drinks on one occasion | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: John Cunningham, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada